CLINICAL TRIAL: NCT05156814
Title: A Prospective, Multicenter, Randomized, Open-label, Comparative Study in Three Parallel Groups to Evaluate the Efficacy and Safety of the Fixed-dose Combination of Estradiol / Dydrogesterone (Femoston® 1 or Femoston® 2, Coated Tablets) and the Combination Therapy of Dydrogesterone (Duphaston®, Coated Tablets) Plus Estradiol (Divigel, Gel for Topical Application, 0.1%) and Monotherapy With Cimicifuga Racemosa Rhizomatum Extract (Klimadynon®) in Perimenopausal Women
Brief Title: Comparative Study to Evaluate the Efficacy and Safety of the Fixed-dose Combination of Estradiol / Dydrogesterone in Perimenopausal Women
Acronym: Violet
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scientific Research Institute of Public Health, Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESDYC001
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Perimenopausal Disorder; Hot Flashes
Keywords: hot flashes; Estradiol; Dydrogesterone; Cimicifuga racemosa; Perimenopausal Women
MeSH Terms: conditions — Hot Flashes | interventions — Dydrogesterone; Klimadynon; Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fixed-dose Combination (FDC) estradiol / dydrogesterone (Experimental): Femoston® 1 (1 mg estradiol / 10 mg dydrogesterone), Femoston® 2 (2 mg estradiol / 10 mg dydrogesterone)
  Interventions: Drug: Femoston® 1, Femoston® 2
- Combination therapy with estradiol and dydrogesterone (Active Comparator): Duphaston®, 10 mg and Divigel, 0.1%
  Interventions: Drug: Duphaston; Drug: Divigel
- non-hormonal therapy (Active Comparator): Cimicifuga racemosa rhizomatum extract (Klimadynon®)
  Interventions: Drug: Klimadynon

INTERVENTIONS:
Drug: Femoston® 1, Femoston® 2 — Femoston® 1 (1 mg estradiol / 10 mg dydrogesterone), Femoston® 2 (2 mg estradiol / 10 mg dydrogesterone)
  Arms: Fixed-dose Combination (FDC) estradiol / dydrogesterone
Drug: Duphaston — Duphaston®, 10 mg
  Arms: Combination therapy with estradiol and dydrogesterone
Drug: Klimadynon — Cimicifuga racemosa rhizomatum extract
  Arms: non-hormonal therapy
Drug: Divigel — Divigel, 0.1%
  Arms: Combination therapy with estradiol and dydrogesterone

SUMMARY:
To obtain new data allowing personalizing continuous hormonal therapy in perimenopausal women in Russia, the following clinical study is going to be conducted in the Russian Federation:

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian women in perimenopause (STRAW -1/ +1a) with an intact uterus.
2. Age from 40 to 55 years old as of the time of screening.
3. Absence of natural menstruations within 4 months, but not longer than for 12 months.
4. 50 or more episodes of "hot flashes" in the last 7 days according to the patient diary (at the screening).
5. Patients scoring more than 12 points on the Greene Scale.
6. Follicle-Stimulating Hormone (FSH) levels more than 25 IU/L, estradiol levels less than 190 pmol/L.
7. Consent to the use of barrier methods of contraception.
8. Body mass index <30 kg / m2.
9. Signed Informed Consent Form.
10. Mammography performed within 6 months prior to inclusion in the study.
11. Absence of clinically significant deviations according to the results of medical examination: physical examination (including assessment of the state of the mammary glands), measurement of indicators of vital body functions (blood pressure, heart rate, respiratory rate and body temperature) and gynecological examination.
12. The patient's consent to perform all research procedures and adhere to all restrictions provided for by the research protocol.

Exclusion Criteria:

1. Smoking.
2. Administration of drugs from the prohibited therapy list.
3. Known hypersensitivity to estradiol, dydrogesterone, to the active component of the drug Klimadynon® (dry extract of rhizomes of cimicifuga racemose) or to any of the excipients of the study drugs.
4. Pregnancy and breastfeeding.
5. Abnormal uterine bleeding from the vagina of unclear etiology within 12 months before the screening stage.
6. Breast cancer (diagnosed, suspected, or past).
7. Estrogen-dependent malignancies of the sex organs, including endometrial cancer (diagnosed, suspected, or past).
8. Known or suspected progestogen-dependent neoplasms (e.g. meningioma).
9. Untreated endometrial hyperplasia.
10. Venous and arterial thrombosis/thromboembolism, currently or in history (including deep vein thrombosis, pulmonary embolism, myocardial infarction, ischemic or hemorrhagic stroke; angina pectoris, transient ischemic attack).
11. Diagnosed hereditary or acquired predisposition to arterial or venous thrombosis/thromboembolism (eg, hyperhomocysteinemia, deficiency of protein C, protein S or antithrombin III, the presence of antiphospholipid antibodies).
12. Acute or chronic liver disease in history (in case of deviation from a norm of liver function indicators); benign and malignant liver tumors (including hemangioma, adenoma, liver cancer) or an increase in Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) activity detected during screening by more than 1.5 times relative to the upper limit of normal.
13. Porphyria.
14. Epilepsy.
15. Brain disorders and traumas.
16. Galactose intolerance, lactase deficiency, glucose-galactose malabsorption syndrome.
17. Cholestatic jaundice and/or severe cholestatic itching (especially during a previous pregnancy or sex hormone intake).
18. Uncontrolled hypertension.
19. Diabetes mellitus.
20. Adenomyosis grade >3 and uterine myoma (more than 3 nodes with an intermuscular or subserous arrangement with a diameter of more than 3 cm) and / or centripetal growth/submucous node location.
21. Cholelithiasis.
22. Systemic lupus erythematosus.
23. Bronchial asthma.
24. Otosclerosis.
25. Known renal or hepatic insufficiency.
26. Ovarian cysts >6 mm based on results of ultrasound scanning.
27. Endometrial thickness ≥5 mm according to transvaginal ultrasound.
28. Migraine headache or a history of severe migraine-type headaches.
29. Other medical conditions which could interfere with the study-related procedures and/or influence the efficacy of the study drug.
30. Simultaneous intake of excluded drugs.
31. Participation in any other clinical study within 3 months before screening.
32. Pathological result of smear for cytology (PAP test) and Human papillomavirus (HPV) test.
33. The use of estrogens or combination drugs for hormone replacement therapy (HRT) within 6 months before the start of the study.
34. Higher risk of thromboembolic complications due to prolonged immobilization for 2 weeks before the screening stage (for example, as a result of trauma or surgery).
35. Previous major surgical interventions (including abdominal) within 6 months before the start of the study.
36. Tumor of the pituitary gland.
37. Severe pathology of the cardiovascular system: complicated lesions of the valvular apparatus of the heart, uncontrolled drug arrhythmia, chronic heart failure I - IV functional class.
38. Sickle cell anemia.
39. Congenital hyperbilirubinemia (Gilbert, Steven-Johnson and Rotor).
40. A history of pancreatitis with severe hypertriglyceridemia.
41. Polyp in the uterine cavity.
42. Use of any drugs in the form of prolonged-release injections or implants within 3 months before the screening stage.
43. A history of any other malignant neoplasms within 5 years prior to the study, with the exception of adequately treated squamous cell skin cancer.
44. Anamnestic data on any clinically significant disease of the kidneys, lungs, gastrointestinal tract, skin and subcutaneous tissues, musculoskeletal system, blood and lymphatic system, nervous system.
45. Positive blood test for HIV, hepatitis B and C, syphilis.
46. Alcoholism, drug addiction in history.
47. Prior endometrial ablation therapy.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Changes in the average number of "hot flashes" per day* as percentages according to data from the patient diary after 84 days (3 cycles) since the initiation of treatment compared to baseline (Visit 0). | 84 days

SECONDARY OUTCOMES:
The change in the total score on the Greene Climacteric Scale at the end of the therapy (364 days) compared to baseline. | 364 days
  This scale includes 21 symptom-questions to assess the emotional-mental state (questions 1-11), somatic manifestations (questions 12 to 18), vasomotor status (questions 19 and 20) and sexual status (21 questions). There are 4 answer options for each question, as in the assessment of the Kupperman index: symptoms do not bother at all - 0 points, slightly bother - 1 point, bother quite strongly - 2 points, extremely pronounced - 3 points. Indicators characteristic of the presence of anxiety or depression - 10 points or more, scored in the first 11 questions. The presence of somatic disorders - 6 or more points in 12-18 questions. Violation of vasomotor function - 4 or more points in 19 and 20 questions.
The frequency of "hot flashes" after 84 days since the initiation of treatment. | 84 days
Changes in the intensity of of menopausal symptoms calculated using the Menopause Rating Scale (MRS) after 84, 168, and 364 days since the treatment initiation compared to baseline (Visit 0). | 84 days, 168 days, 364 days
  The questionnaire has 11 items and option to check one of 5 degrees of severity of symptoms (from 0 (none) to 5 (very severe) points at the questionnaire).
Changes according to the Greene Climacteric Scale in each of the 4 subscales after 84, 168, and 364 days since the initiation of treatment compared to baseline (Visit 0). | 84 days, 168 days, 364 days
  This scale includes 21 symptom-questions to assess the emotional-mental state (questions 1-11), somatic manifestations (questions 12 to 18), vasomotor status (questions 19 and 20) and sexual status (21 questions). There are 4 answer options for each question, as in the assessment of the Kupperman index: symptoms do not bother at all - 0 points, slightly bother - 1 point, bother quite strongly - 2 points, extremely pronounced - 3 points. Indicators characteristic of the presence of anxiety or depression - 10 points or more, scored in the first 11 questions. The presence of somatic disorders - 6 or more points in 12-18 questions. Violation of vasomotor function - 4 or more points in 19 and 20 questions.
Changes according to the "Hot Flush" Related Daily Interference Scale (HFRDIS) after 84, 168, and 364 days since the initiation of treatment compared to baseline (Visit 0). | 84 days, 168 days, 364 days
  The HFRDIS is 10-item scale measuring the degree hot flashes interfere with nine daily activities.
The average treatment satisfaction score according to the Likert Scale after 84, 168, and 364 days since the initiation of treatment. | 84 days, 168 days, 364 days
  Assessment of satisfaction with treatment is based on the patient's assessment of the degree of his consent or disagreement with the statements in a hierarchical sequence from "completely disagree" through "disagree", "find it difficult to answer", "agree" to "completely agree".
Changes in the adipose tissue according to densitometry results after 364 days of treatment compared to baseline (Visit 0). | 364 days
Changes in the waist circumference after 364 days of treatment compared to baseline (Visit 0). | 364 days
Changes in the bone tissue according to densitometry results after 364 days of treatment compared to baseline (Visit 0). | 364 days
Changes in the bone resorption marker β-Cross laps after 364 days of treatment compared to baseline (Visit 0). | 364 days
Changes in the bone formation marker (P1NP) after 364 days of treatment compared to baseline (Visit 0). | 364 days

CONTACTS AND LOCATIONS:
Locations (1):
- Federal State Budget Institution "National Medical Research Center for Obstetrics, Gynecology and Perinatology named after Academician V.I.Kulakov", Moscow, Russia